CLINICAL TRIAL: NCT01953172
Title: Exploratory, Double-blind, Randomized, Placebo Controlled Study of AMP-886 in the Elderly
Brief Title: Health Status and Quality of Life in the Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Unilever R&D (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: FDS-NBU-1034
Record Dates: First submitted 2013-09-13; First posted 2013-09-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Quality of Life
MeSH Terms: interventions — tocotrienol, alpha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo capsules (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo
- AMP-886 (alpha-tocotrienol) in capsules (Experimental): AMP-886 (alpha-tocotrienol) in capsules
  Interventions: Dietary Supplement: AMP-886

INTERVENTIONS:
Dietary Supplement: AMP-886 — AMP886 (alpha-tocotrienol) encapsulated in gelatin capsules
  Other Names: alpha-tocotrienol
  Arms: AMP-886 (alpha-tocotrienol) in capsules
Other: Placebo — Placebo
  Arms: Placebo capsules

SUMMARY:
The study is designed to investigate the effect of AMP886 (alpha-tocotrienol) on health status and quality of life measures, cognitive functioning, oxidative stress, inflammation markers and other symptoms effects on skin, sleep and vision in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 65-85 years old
* ECOG Performance score 0 to 1
* Body mass index 22-30 kg/m2
* Body weight >60 kg
* Habit to consume standard breakfast like toast, bread, butter/margarine, eggs, bacon, cereals with milk
* Comply with protocol and likely to be compliant with prescribed product

Exclusion Criteria:

* Renal insufficiency or failure at screening
* Current or previous positive documented history of any chronic inflammatory state including chronic infection, arthritis, or collagen vascular disorder.
* Comorbid medical conditions
* Use of prescription medication for chronic conditions
* Use of hormone replacement therapy (with the exception of levothyroxine)
* Uncontrolled hypertension
* Use of hemostatic agents
* Hemorrhagic disorder and/or coagulation disorder
* Clinically important bleeding within 90 days prior to screening visit
* Fat malabsorption syndromes
* Constipation and/or abdominal pain/discomfort that require dietary supplements or medical therapy
* History of smoking within 1 year prior to visit 1.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on health status
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on quality of life measures
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on cognitive functioning
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on oxidative stress
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on inflammation markers
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on skin
Effects on health status and quality of life | up to 24 weeks
  Objective of this exploratory study is to evaluate the effects of AMP886 on vision

CONTACTS AND LOCATIONS:
Overall Officials: C Verhoeven, PhD, Study Director — Unilever Research and Development
Locations (3):
- United Kingdom (3):
  - Whipps Cross Hospital, London
  - King's College Hospital, London
  - Central Manchester Hospital, Manchester